CLINICAL TRIAL: NCT04795076
Title: Effect of Feeding With Nutrient Dense Formula Compared to Standard Formula on Anthropometric Indices, in Malnourished Infants and Children With Congenital Heart Defects After Repair Surgery
Brief Title: Effect of Feeding With Nutrient Dense Formula in Malnourished Infants and Children With Congenital Heart Defects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shahid Beheshti University (Other)
Responsible Party: Principal Investigator, Javad Nasrollahzadeh, Associate Professor, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 22213
Record Dates: First submitted 2021-03-06; First posted 2021-03-12 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-02

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Infant Formula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard formula (Placebo Comparator): Feeding the infant or child with the regular formula which is prepared with standard concentrations
  Interventions: Dietary Supplement: Infant formula
- Nutrient-dense formula (Active Comparator): Feeding the infant or child with the nutrient-dense formula which is prepared by concentrating regular formula.
  Interventions: Dietary Supplement: Infant formula

INTERVENTIONS:
Dietary Supplement: Infant formula — Regular infant formula will be concentrated to give a calorie density of about 90 kcal/100 mL.

SUMMARY:
Infants with congenital heart disease (CHD) are usually born with a normal weight but develop malnutrition over time, and about 20-50% of these children are usually malnourished. Malnutrition in these patients is multifactorial. To compensate for the increased need for infants and children with CHD, an increase in their caloric intake has been suggested. However, these patients may not be able to receive enough to meet the increased needs and catch-up growth. One of the suggested solutions in these patients to compensate for inadequate food intake is to increase the caloric density of milk or formula. For this purpose, the use of special formulas with higher calorie density or enrichment of normal formula or breast milk using special enrichment formula could be suggested. In the present study, the effect of increasing calorie intake by increasing the concentration of normal formula in comparison with formula with standard concentration on weight gain and other anthropometric indices of CHD patients with malnutrition will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Infant and children 6 to 24 months with CHD undergoing repair surgery
* Malnutrition (weight for age Z score ≤ -1)

Exclusion Criteria:

* Allergy to cow's milk protein
* Preterm infant or infant weighing less than 2500 grams at birth
* Children with chromosomal disease (Down, Turner)

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 65 (Actual)
Dates: Start 2021-04-03 (Actual); Primary Completion 2022-02-09 (Actual); Study Completion 2022-02-09 (Actual)

PRIMARY OUTCOMES:
Weight | Change from baseline at 2 months
  Body weight of infant or child

SECONDARY OUTCOMES:
Length | Change from baseline at 2 months
  Recumbent length of infant or child
Mid-arm circumference | Change from baseline at 2 months
  mid upper-arm circumference of infant or child
Head circumference | Change from baseline at 2 months
  Head circumference
IGF1 | Change from baseline at 2 months
  Serum IGF1

CONTACTS AND LOCATIONS:
Locations (1):
- Rajaei Cardiovascular, Medical & Research Center, Tehran, Iran

IPD SHARING:
Plan to Share IPD: Undecided